CLINICAL TRIAL: NCT06618820
Title: Randomized Control Trial for Oral Extended Tranexamic Acid After Total Knee Arthroplasty
Brief Title: Extended Oral Tranexamic Acid After Total Knee Arthroplasty
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, Chris Holland, MD, Instructor, Department of Orthopaedic Surgery and Biomechanical Engineering, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-10171-FB
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Osteo Arthritis Knee; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Tranexamic Acid; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to randomization assignment until completion of their one year follow up visits. The care provider, investigators and outcome assessor will be blinded to randomization assignment until completion of data analysis. The investigators and care providers will not be blinded to randomization assignment if an adverse event occurs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Patients will receive 10 doses of microcrystalline cellulose (3 capsules per dose) from postoperative day (POD) 1 to POD 10.
  Interventions: Drug: Placebo
- 3-day tranexamic acid (TXA) (Experimental): Patients will receive three 1950 milligram (mg) doses of Oral TXA (three 650mg capsules per dose) from POD 1 to POD 3 and 7 doses of Placebo from POD 4 to POD 10.
  Interventions: Drug: Tranexamic acid; Drug: Placebo
- 10-day TXA (Experimental): Patients will receive ten 1950mg doses of Oral TXA (three 650mg capsules per dose) from POD 1 to POD 10.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — One dose consists of three 650 milligram (mg) capsules, to be taken orally.
  Arms: 10-day TXA; 3-day tranexamic acid (TXA)
Drug: Placebo — One dose consists of three microcrystalline cellulose capsules.
  Other Names: microcrystalline cellulose
  Arms: 3-day tranexamic acid (TXA); Placebo

SUMMARY:
The utilization of intraoperative tranexamic acid (TXA), whether administered intravenously or orally, has become a standard practice in total joint arthroplasty (TJA). Multiple studies have demonstrated the positive impact that TXA application has on clinical outcomes, including decreased blood loss and transfusion rates, decreased early swelling and ecchymosis, improved early recovery, and potentially superior long-term outcomes. Its ability to mitigate risk of blood loss made ambulatory total knee arthroplasty (TKA) safer for patients. The safety of intraoperative TXA use has also been documented. Sabbag et al. showed that TXA does not increase the risk of venous thromboembolism (VTE), even in those patients who are deemed high-risk. Multiple routes of TXA administration have been studied with each route demonstrating effectiveness in reducing blood loss. Findings showed that oral TXA is noninferior to intravenous TXA, though the median time to reach a target concentration is longer via the oral route and bioavailability is lower. With the benefits of intraoperative TXA clearly documented in literature, multiple centers investigated the utilization of extended TXA postoperatively in hopes of enhancing patient safety and reducing length of stay and healthcare cost. However, these studies reported conflicting outcomes and mostly focused on estimated blood loss, instead of patient reported outcomes.

The purpose of this study is to assess the effectiveness and safety of a varying extended oral TXA regimen during the postoperative period. Further, the investigators aim to determine the optimal duration of the TXA regimen to maximize its impact. The investigators hypothesize that an extended oral TXA regimen is safe and effective in improving clinical outcomes in TKA patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older.
2. Primary TKA at a Campbell Clinic Surgery Center, with implant at the discretion of the treating surgeon.
3. Willing to participate in the study.
4. Fluent in oral and written English.

Exclusion Criteria:

1. Revision TKA.
2. Preoperative use of anticoagulants (81mg aspirin is allowed).
3. Prior history of deep vein thrombosis.
4. Prior history of cancer (with the exception of non-melanoma/metastatic skin cancers, low-grade non-metastatic benign soft tissue tumors, thyroid cancers and low grade, non-metastatic prostate cancers).
5. Known allergy or hypersensitivity to TXA.
6. Patients who are using combination hormonal contraception.
7. History of seizure disorder.
8. History of adult onset colorblindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Forgotten Joint Score - Knee | Enrollment; 2-week postoperative; 6-week postoperative; 12-week postoperative; 1-year postoperative.
  The Forgotten Joint Score measures how much the patient is aware of their affected knee during activities of daily living. A score of 0 indicates that the patient is always aware of their affected knee whereas a score of 100 indicates that the patient is not aware of their affected knee during activities of daily living.
Range of Motion | Enrollment; 2-week postoperative; 6-week postoperative; 12-week postoperative; 1-year postoperative.
  Passive flexion and extension range of motion of the surgical knee will be assessed with a goniometer in degrees.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement | Enrollment; 2-week postoperative; 6-week postoperative; 12-week postoperative; 1-year postoperative.
  This questionnaire assesses patients' knee health with 0 representing total disability and 100 represents perfect knee health.
Patient-Reported Outcomes Measurement Information System | Enrollment; 2-week postoperative; 6-week postoperative; 12-week postoperative; 1-year postoperative.
  This questionnaire assesses patients' overall health and wellbeing with a T-score of 16.2 representing most severe physical impairment and a T-score of 67.7 represents best possible state of health.
Visual Analog Scale | Enrollment; postoperative day 1 to postoperative day 14; 2-week postoperative; 6-week postoperative; 12-week postoperative; 1-year postoperative.
  This questionnaire assesses patient's pain level with 0 being no pain at all and 10 being worst pain possible.
Opiate pill count | postoperative day 1 to postoperative day 14; 2-week postoperative; 6-week postoperative; 12-week postoperative; 1-year postoperative.
  The investigators will record the number of opiate medication taken by the patient and calculate morphine milligram equivalents.
Ambulatory aid | Enrollment; postoperative day 1 to postoperative day 14; 2-week postoperative; 6-week postoperative; 12-week postoperative; 1-year postoperative.
  The investigators will record the use of ambulatory aid, such as walker.
Adverse Event | From signing consent form to completion of 1 year follow up visit.
  The investigators will monitor for adverse events, including but not limited to deep venous thrombosis, and pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Holland, MD, MS, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Germantown, Tennessee, United States